CLINICAL TRIAL: NCT06352931
Title: Transcranial Ultrasound and Transcranial Doppler in Diagnosis and Detection of Outcome in Infants With Neurological Diseases
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Sami Abdelrahman Khalifa, assistant lecturer, Assiut University
Other Study IDs: TCD & TCUS in infants
Record Dates: First submitted 2024-04-03; First posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: Trancranial Doppler

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: transcranial and transcranial dopp;er — All patients will be subjected to Transcranial ultrasound examination and compared with other neuroimaging modalities: CT brain or MRI brain and/or MRA & MRV.
  Patients suspected to have ischemic or hemorrhagic disorder, CNS infection or increase intracranial pressure will be evaluated with transcranial Doppler ultrasound and compared with other neuroimaging modalities.

SUMMARY:
To evaluate the accuracy of transcranial ultrasound in detection of brain pathology in infants with neurological diseases and value of transcranial Doppler in evaluation of intracerebral blood flow in comparison with other radiological modalities according to available imaging.

DETAILED DESCRIPTION:
Neurologic disorders are seen commonly in children, especially in developing countries [1]. They significantly contribute to morbidity and disability in children and contribute significantly to chronic illness and its burden on children [2]. They can result from genetic or environmental factors or a combination of both [3]. Many relatively rare conditions which have high mortality in the past, like cancers, spinal bifida, and sickle cell anemia, now survive and contribute to the burden of chronic childhood diseases [4]. That's why early detection and management of neurological manifestations is very important.

Head and neck radiology has evolved during the century since the discovery of the x ray in 1895 by Wilhelm Conrad Roentgen. In the first few decades, conventional radiography was the diagnostic modality for evaluation of head and neck diseases, Linear tomography was further enhanced with the introduction of thin-section polytomography especially of the temporal bone in 1954, Computed tomography in 1972 and magnetic resonance imaging in 1982 improved our diagnostic capabilities by enabling location and characterization of tumors, cysts, and inflammatory processes in the head and neck and aiding in earlier diagnosis and treatment (5) Dewbury et al in 1980 first reported the use of anterior fontanelle as a bone free window through which brain can be imaged. Since then this technique has become widely accepted and is regarded as the primary imaging method for the neonatal brain [6] A cranial ultrasound is also known as a 'head scan'. Sound waves are used to look at the brain structure and the fluid spaces within the brain (ventricles). It does not involve any ionizing radiation [7] .

Ultrasound waves travel into tissue and are reflected back to the probe at a rate determined by the target tissue's consistency. Reflections of sound that return to the probe are called echoes and are determined by two different materials' interfaces.[8] Cranial US has become an essential primary diagnostic screening tool for intracranial pathologic conditions in infants. Significant technical advances including use of high frequency transducers, imaging through secondary acoustic windows, and incorporation of Doppler imaging allow a comprehensive evaluation of the brain. In addition, US is noninvasive, requires no sedation, can be performed at the bedside with minimal disturbance to the neonate and infants, and may be repeated as often as necessary. [9] Various studies have demonstrated high sensitivity and specificity of transcranial ultrasound in detection of various intracranial abnormalities [10].

Most cranial sonographic examinations are performed in coronal and the sagittal planes, through the anterior fontanelle that remains useful for scanning 12-14 months of age infants . Posterior and mastoid fontanelles provide a better window for evaluation of posterior fossa structures Pterion is an important window for evaluation of circle of willis .[11] In spite of these views are indispensable for evaluation of posterior fossa malformations as they provide highly detailed views of the cerebellum, fourth ventricle, cisterna magna, and upper spinal canal. Coronal and sagittal planes are the most useful imaging planes for cranial sonography and allow a comprehensive brain examination, they afford a useful window for a limited age only i.e. up to 6 months. [12] Transcranial ultrasound helps in imaging of brain and intraventricular chambers through sound waves reflected from the brain and cerebrospinal fluid (CSF). For the evaluation of extra-axial fluid space, meninges, sinuses, convolutional markings and cerebral cortex, high frequency linear array transducers are better to be used .[13] Many pathological lesions could be detected by trans-cranial ultrasound as Neonatal hypoxic lesions and intracranial hemorrhagic lesions with the resulting ventricular dilatation. Also, it is the technique of choice in detection of periventricular leukomalecia (PVL) . It can detect many congenital malformations of the brain as hydrocephalus secondary to aqueductal stenosis, Chiari II malformation, posterior fossa cystic abnormalities including Dandy-Walker spectrum, holoprosencephaly , schizencephaly, agenesis of the corpus callosum (CC), vein of Galen malformation and arachnoid cysts. Cranial ultrasound also shows high sensitivity in detection of calcification foci resulting from congenital TORCH infection. Finally Intracranial neoplasms which are rare in neonates and infants can be seen by cranial sonography [14].

Transcranial Doppler (TCD) ultrasound including color flow(CF) and pulsed wave (PW) enables the bedside evaluation of these patients; it is a non-invasive, readily available technique for the real-time assessment and monitoring of cerebral blood flow. TCD shows high sensitivity and specificity for the diagnosis of vasospasm after subarachnoid hemorrhage, acute middle cerebral artery (MCA) occlusions and brain death [15]. Furthermore, TCD is a reliable method for estimating the intracranial pressure (ICP) - particularly in the context of traumatic brain injury [16]. The use of TCD has also been described in the management of sepsis [17], central nervous system (CNS) infections [18], and liver and kidney failure [19,20] , there is good evidence to support the use of TCD in screening for sickle cell disease in children and whose risk of a first stroke would be reduced by a blood transfusion [21] Three key parameters can be obtained from the Doppler spectrum: flow direction, velocities, and indices for arterial resistance. Flow direction can be assessed by the colour code. By convention, flow towards the transducer is coded in red and is plotted above the baseline in the pulsed wave Doppler-spectrum; flow away from the transducer is coded in blue and plotted below the baseline. The most commonly used velocity parameter is the time average mean of the maximal velocities (TAMX), also called mean velocity, obtained by manual or automated outlining of the envelope of the spectral waveform over one cardiac cycle. The peak systolic velocity (PSV) and end diastolic velocity (EDV) can also be measured. Two indices reflecting the downstream vascular resistance can be calculated. The pulsatility index (PI) is calculated as PI = (PSV -EDV) / TAMX. The resistance index, RI, is equal to (PSV - EDV) / PSV. [22].

ELIGIBILITY:
Inclusion Criteria:

Newborns and infants (from birth to 2years) with open anterior fontanelle presented with any neurological signs e.g: convulsions, disturbed conscious level &coma, suspected CNS infection macrocephaly, head trauma, multiple congenital anomalies, persistent vomiting, bulging anterior fontanelle, developmental delay, neurological deficit.

-

Exclusion Criteria:

1-Children with closed anterior fontanelle. 2- Infants without neurological signs.

-

Ages: 1 Day to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Newborns and infants (from birth to 2years) with open anterior fontanelle presented with any neurological signs e.g: convulsions, disturbed conscious level &coma, suspected CNS infection macrocephaly, head trauma, multiple congenital anomalies, persistent vomiting, bulging anterior fontanelle, developmental delay, neurological deficit
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
To evaluate the accuracy of transcranial ultrasound in detection of brain pathology in infants with neurological diseases and value of transcranial doppler | one year duration
  To evaluate the accuracy of transcranial ultrasound in detection of brain pathology in infants with neurological diseases and value of transcranial Doppler in evaluation of intracerebral blood flow in comparison with other radiological modalities according to available imaging.

REFERENCES:
- [Background] Kawakatsu Y, Kaneko S, Karama M, Honda S. Prevalence and risk factors of neurological impairment among children aged 6-9 years: from population based cross sectional study in western Kenya. BMC Pediatr. 2012 Dec 3;12:186. doi: 10.1186/1471-2431-12-186. PMID 23206271
- [Background] Weber AL. History of head and neck radiology: past, present, and future. Radiology. 2001 Jan;218(1):15-24. doi: 10.1148/radiology.218.1.r01ja2715. PMID 11152774
- [Background] Richer EJ, Riedesel EL, Linam LE. Review of Neonatal and Infant Cranial US. Radiographics. 2021 Nov-Dec;41(7):E206-E207. doi: 10.1148/rg.2021210089. No abstract available. PMID 34723697
- [Background] Gupta P, Sodhi KS, Saxena AK, Khandelwal N, Singhi P. Neonatal cranial sonography: A concise review for clinicians. J Pediatr Neurosci. 2016 Jan-Mar;11(1):7-13. doi: 10.4103/1817-1745.181261. PMID 27195026